CLINICAL TRIAL: NCT04028895
Title: Assessement of the Diagnostic Interest in Insulin Resistance of the Specific and Quantitative ELISA Assay of a Plasma Biomarker of Cellular Glucose Capture: the Secreted IRAP Protein (Regulated Amino Peptidase Insulin)
Brief Title: Diagnostic Interest of the IRAP Protein (Insulin Regulated Amino Peptidase) in Insulin Resistance
Acronym: IRAP-IR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: stopped by the sponsor
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC18.326
Record Dates: First submitted 2019-05-23; First posted 2019-07-23 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Insulin Resistance Syndrome
Keywords: IRAP; Insulin Regulated Amino Peptidase
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Other)
  Interventions: Diagnostic Test: Dosage of IRAP during OGTT

INTERVENTIONS:
Diagnostic Test: Dosage of IRAP during OGTT — Visit 1: oral glucose tolerance test. visit 2: hyperinsulinemic euglycemic clamp

SUMMARY:
There is currently no reliable, diagnostic tests of insulin resistance other than the hyperinsulinemic euglycemic clamp which, due to its constraints and cost, is reserved for research. The insulin-Regulated aminopeptidase (IRAP) protein is a direct marker of insulin-dependent glucose cell capture and thus it blood concentration seems to be a good diagnostic test of insulin resistance.

The purpose of this study is to assess a plasma essay of IRAP protein for evaluation of insulin resistance during an oral glucose tolerance test (OGTT).

DETAILED DESCRIPTION:
This study consists of two visits, from three to fifteen days apart. Patients with different levels of insulin resistance will be enrolled in this study.

The level of insulin resistance will be estimated with a hyperinsulinemic euglycemic clamp that will be performed at the second visit.

The first visit :

* Subjects will be on an empty stomach
* A blood test including HbA1C, C-Peptid, lipid profile, creatinine,urea, hepatic workup
* An oral glucose tolerance test (OGTT) of 3 hours will be performed. Blood samples will be taken two time (T-15', T0) 15 minutes apart at Baseline (before taking the glucose). And then after the glucose intake, blood sample will be taken every 15 minutes (T15', T30', T 45', T60', T75', T90', T105', T120' and 180') to measure insulinemia, blood sugar, and IRAP concentration.

The second visit includes a 3-hours hyperinsulinemic euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* Patient without known diabetes
* Abdominal perimeter greater than 80 cm for women and greater than 94 cm for men
* Patient affiliated to social security insurance or beneficiary of social security insurance.
* Signed consent

Exclusion Criteria:

* Consumption of narcotic
* Medication that may interfere with glucose metabolism
* History of bariatric surgery
* Known acute or chronic renal insufficiency
* Hyperinsulinemic euglycemic clamp contraindication
* Contraindications with insulin, G20 glucose and Di-potassium phosphate
* Histories of coronary pathology
* History of heart rhythm disorders requiring chronic treatment
* Period of fast
* Pregnant women

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
IRAP concentration during OGTT. | At the first visit (Day 0)
  The level of insulin resistance will be estimated with a hyperinsulinemic euglycemic clamp. The specificity and sensitivity of the IRAP concentration for the diagnosis of insulin resistance will be determined at every time of the OGTT.

SECONDARY OUTCOMES:
Kinetic profile of IRAP concentration in 3-hours OGTT | At the first visit (Day 0)
  Evolution of the concentration of IRAP at each point of the OGTT.
Diagnostic value of IRAP | At the first visit (Day 0)
  Comparison of AUC (area under curve) of IRAP's ROC curves with that of insulin.
Diagnostic value of IRAP | At the first visit (Day 0)
  Comparison of AUC (area under curve) of IRAP's ROC curves with that of glucose.
Diagnostic value of IRAP | At the first visit (Day 0)
  Comparison of AUC (area under curve) of IRAP's ROC curves with that of resistance indexes.
Diagnostic value of the concentration of other biomarkers (not yet determined) | During the first visit (Day 0)
  The diagnostic value of other potential insulin resistance biomarkers will be tested using the same methodology as for IRAP.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Service de Nutrition clinique et CRNH Auvergne, Clermont-Ferrand
  - Inserm CIC1406, clinical research center, Grenoble Alpes university hospital, Grenoble
  - CRNH Rhône-Alpes et Centre Hospitalier LYON Sud, Lyon
  - Endocrinologie-Diabétologie-Nutrition et CIC, CHU DE MONTPELLIER, Montpellier